CLINICAL TRIAL: NCT02455245
Title: A Phase III Study Comparing Two Carboplatin Containing Regimens for Children and Young Adults With Previously Untreated Low Grade Glioma
Brief Title: A Study Comparing Two Carboplatin Containing Regimens for Children and Young Adults With Previously Untreated Low Grade Glioma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alicia Lenzen (Other)
Responsible Party: Sponsor-Investigator, Alicia Lenzen, Attending, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LGG 14C03
Record Dates: First submitted 2015-04-13; First posted 2015-05-27 (Estimated); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Low Grade Glioma
MeSH Terms: interventions — Carboplatin; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Carboplatine and Vincristine (Active Comparator): Induction: 10 weeks of Carboplatin and Vincristine therapy. Carboplatin 175 mg/m2 give an an IV infusion weeks 1, 2, 3, 4, 7, 8, 9, 10. Vincristine 1.5mg/m2 (0.05 mg/kg if child less than 12 kg) (maximum dose 2.0 mg) give as an IV bolus infusion on weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10.
  Maintenance: Maintenance consists of 8, 6-week cycles of chemotherapy. It begins week 12 of Induction or when peripheral counts recover with ANC >1,000/µL and platelet count >100,000/µL. Each cycle will consist of 4 weekly doses of carboplatin, three weekly doses of vincristine (given concomitantly with the first 3 weeks of carboplatin), followed by two weeks of rest for a total of 6 weeks. Maintenance will continue for a total of 8 cycles.
  Carboplatin 175 mg/m2 as an IV continuous infusion over 60 minutes on Week 1, 2, 3, 4 of each cycle. Vincristine 1.5 mg/m2 (0.05 mg/ kg for children <12 kg) (maximum dose 2.0 mg) IV bolus infusion on Week 1, 2, 3 of each cycle.
  Interventions: Drug: Carboplatin and Vincristine; Drug: Carboplatin
- Carboplatin alone (Experimental): Carboplatin is given once every four weeks, Each 4-week period is considered a cycle. Regimen B will last for 13 cycles which is equivalent to one year (52 weeks).
  Carboplatin 560 mg/m2 (or 19 mg/kg for children weighing less than 12 kg) IV over 1 hour every 4 weeks
  Interventions: Drug: Carboplatin and Vincristine

INTERVENTIONS:
Drug: Carboplatin and Vincristine — Carboplatin 175 mg/m2 IV infusion Vincristine 1.5mg/m2 IV
Drug: Carboplatin — Carboplatin 560 mg/m2 (or 19 mg/kg for children weighing less than 12 kg) IV
  Arms: Carboplatine and Vincristine

SUMMARY:
This study is trying to learn and understand if the chemotherapy drug called carboplatin works as well as the standard therapy. The standard therapy for Low Grade Glioma (LGG) in children and young adults is using a combination of carboplatin and vincristine. Studies in children have shown that the use of carboplatin alone has promise of being just as effective for treating LGG as standard therapy. Additionally, this study will try to understand if treatment with carboplatin alone is associated with an improved quality of life for LGG patients and their families.

DETAILED DESCRIPTION:
Low grade gliomas are the most common central nervous system (CNS) tumors in the pediatric population. They consist of a heterogeneous group of tumors that are classified as World Health Organization (WHO) grade I or II. This includes astrocytic, oligodendroglial, neuronal and mixed glial- neuronal tumors. The clinical behavior of these tumors varies according to location and histology. The cerebellum is the most common location for low grade gliomas, but they can also arise in the cerebrum, deep midline structures such as the hypothalamus, optic pathway and, less frequently, in the brainstem.

Although the etiology of most childhood LGG is unknown, patients with Neurofibromatosis type 1 (NF-1) are one rare group predisposed to developing CNS tumors. NF-1 is an inherited disorder that affects the nervous system, eyes and skin. In addition, children are at an increased risk for developing optic pathway and hypothalamic low grade gliomas. Fifteen to-20% of NF-1 patients will develop these tumors, and they account for up to 70% of the tumors seen in this location. In half of patients with NF-1 and an optic pathway tumor, the patients are not symptomatic and the mass is found incidentally. Many optic gliomas in NF-1 patients follow an indolent course and stabilize without intervention. Patients are most commonly treated when there is deterioration in their vision or a symptomatic increase in the tumor size. Although the event free survival (EFS) has been reported to be similar between NF1 and non-NF1 patients, overall survival is higher in NF1 patients.

Location, as it affects the extent of surgical resection, plays a key role in the prognosis of all patients with low grade gliomas. Complete surgical resection offers a 90% survival rate at 10 years with often no need for adjuvant chemotherapy or radiation. Unfortunately, a gross total resection is not always possible due to the location of the tumor and its proximity to vital structures in the brain. In patients with an incomplete resection, the 10 year EFS is up to 74% with radiation treatment. However, toxicity from radiation, especially in young children, is significant and includes neurocognitive delays, endocrinopathies, secondary malignancy, ototoxicity and vasculopathy. Therefore, most experts agree that the standard of care in young children is to treat low grade gliomas that require adjuvant therapy after surgical resection/biopsy, or whose tumors are not surgically resectable with chemotherapy first, in order to delay or avoid radiation. This is especially true in children with NF-1, where the risk of a secondary malignancy after radiation therapy can be as high as 50% in the lifetime of the child.

ELIGIBILITY:
Inclusion Criteria:

* Tumor Diagnosis: Low grade gliomas
* Patients must be less than 21 years of age at study entry.
* Central nervous system tumor. Patients with primary spinal cord lesions. Patients with metastatic disease are also allowed.
* No previous therapy for the tumor with the exception of corticosteroids and surgery.
* Performance status:Karnofsky Performance Scale (KPS for > 16 yrs of age) or Lansky Performance Score (LPS for ≤ 16 years of age) ≥ 50 assessed within two weeks prior to registration
* Seizure disorder should be well controlled.
* Normal organ and marrow function
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients who have menstruated and are of childbearing potential must have a negative serum or urine pregnancy test prior to enrollment.
* Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study and for 6 months after the last drug administration.
* Ability of subject or parent/guardian to understand and the willingness to sign a written informed consent/assent document. Informed consent/assent must be signed prior to registration on this study.
* Tissue blocks or slides must be sent. If tissue is unavailable, the study chair must be notified prior to enrollment.

Exclusion Criteria:

* Patients who are receiving any other investigational or chemotherapeutic agents will be excluded.
* Patients with known inability to return for follow-up visits or obtain follow-up studies required to assess for toxicity to therapy.
* Patients with Subepenydmal Giant Cell Astrocytomas are excluded. Patients with intrinsic brainstem tumors of the pons will be excluded from the study.
* History of hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to platinum based chemotherapy.
* Patients with uncontrolled inter-current illness are excluded.
* Females who are pregnant or breast feeding are excluded.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  To compare the progression-free survival (PFS) in patients with previously untreated LGG among patients with and without NF1 utilizing carboplatin/vincristine (standard of care) vs single agent carboplatin (research).

SECONDARY OUTCOMES:
Number of participants who experience improved quality of life as assessed by a Quality of Life questionnaire. | week-6, week-12, month-6, month-12
  To compare the QOL among both regimens.
Tumor response rate of each regimen, assessed by magnetic resonance imaging (MRI) | 3 years
  To estimate tumor response rates of each regimen.
Number of participants who experience toxicity on each regimen | 3 years
  To determine toxicity of each regimen
Number of B-Raf proto-oncogene, serine/threonine kinase (BRAF) mutations that have an association with clinical outcomes. | 3 years
  To assess the molecular findings and correlate with clinical outcome.
Number of aberrations found through whole exome and ribonucleic acid (RNA) sequencing that coordinate with a clinical outcome. | 3 years
  To assess the molecular findings and correlate with clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Lenzen, MD, Principal Investigator — Attending
Locations (21):
- United States (21):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Rady Children's Hospital, San Diego, California
  - Yale University, New Haven, Connecticut
  - Orlando Health, Inc., Orlando, Florida
  - Ann & Robert H. Lurie Children's Hosptial of Chicago, Chicago, Illinois
  - St. Vincent Peyton Manning Children's Hospital, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Saint Louis University at SSM Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Duke University Medical School, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - American Family Children's Hospital, Madison, Wisconsin
  - Medical College of Wiscosin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Sievert AJ, Fisher MJ. Pediatric low-grade gliomas. J Child Neurol. 2009 Nov;24(11):1397-408. doi: 10.1177/0883073809342005. PMID 19841428
- [Background] Gururangan S, Cavazos CM, Ashley D, Herndon JE 2nd, Bruggers CS, Moghrabi A, Scarcella DL, Watral M, Tourt-Uhlig S, Reardon D, Friedman HS. Phase II study of carboplatin in children with progressive low-grade gliomas. J Clin Oncol. 2002 Jul 1;20(13):2951-8. doi: 10.1200/JCO.2002.12.008. PMID 12089224
- [Background] Sharif S, Ferner R, Birch JM, Gillespie JE, Gattamaneni HR, Baser ME, Evans DG. Second primary tumors in neurofibromatosis 1 patients treated for optic glioma: substantial risks after radiotherapy. J Clin Oncol. 2006 Jun 1;24(16):2570-5. doi: 10.1200/JCO.2005.03.8349. PMID 16735710
- [Background] Petronio J, Edwards MS, Prados M, Freyberger S, Rabbitt J, Silver P, Levin VA. Management of chiasmal and hypothalamic gliomas of infancy and childhood with chemotherapy. J Neurosurg. 1991 May;74(5):701-8. doi: 10.3171/jns.1991.74.5.0701. PMID 1901597
- [Background] Packer RJ, Lange B, Ater J, Nicholson HS, Allen J, Walker R, Prados M, Jakacki R, Reaman G, Needles MN, et al. Carboplatin and vincristine for recurrent and newly diagnosed low-grade gliomas of childhood. J Clin Oncol. 1993 May;11(5):850-6. doi: 10.1200/JCO.1993.11.5.850. PMID 8487049
- [Background] Lafay-Cousin L, Sung L, Carret AS, Hukin J, Wilson B, Johnston DL, Zelcer S, Silva M, Odame I, Mpofu C, Strother D, Bouffet E. Carboplatin hypersensitivity reaction in pediatric patients with low-grade glioma: a Canadian Pediatric Brain Tumor Consortium experience. Cancer. 2008 Feb 15;112(4):892-9. doi: 10.1002/cncr.23249. PMID 18098210
- [Background] Korinthenberg R, Neuburger D, Nikkhah G, Teske C, Schnabel K, Calaminus G. Assessing quality of life in long-term survivors after (1)(2)(5)I brachytherapy for low-grade glioma in childhood. Neuropediatrics. 2011 Jun;42(3):110-5. doi: 10.1055/s-0031-1283111. Epub 2011 Jul 7. PMID 21739406
- [Background] Bryant R. Managing side effects of childhood cancer treatment. J Pediatr Nurs. 2003 Apr;18(2):113-25. doi: 10.1053/jpdn.2003.11. PMID 12720208
- [Background] Woodgate RL, Degner LF, Yanofsky R. A different perspective to approaching cancer symptoms in children. J Pain Symptom Manage. 2003 Sep;26(3):800-17. doi: 10.1016/s0885-3924(03)00285-9. PMID 12967729
- [Background] Kazak AE, Simms S, Rourke MT. Family systems practice in pediatric psychology. J Pediatr Psychol. 2002 Mar;27(2):133-43. doi: 10.1093/jpepsy/27.2.133. PMID 11821497
- [Background] Mulhern RK, Carpentieri S, Shema S, Stone P, Fairclough D. Factors associated with social and behavioral problems among children recently diagnosed with brain tumor. J Pediatr Psychol. 1993 Jun;18(3):339-50. doi: 10.1093/jpepsy/18.3.339. PMID 8340843
- [Background] Katz ER, Varni JW. Social support and social cognitive problem-solving in children with newly diagnosed cancer. Cancer. 1993 May 15;71(10 Suppl):3314-9. doi: 10.1002/1097-0142(19930515)71:10+3.0.co;2-1. PMID 8490874
- [Background] O'Malley JE, Koocher G, Foster D, Slavin L. Psychiatric sequelae of surviving childhood cancer. Am J Orthopsychiatry. 1979 Oct;49(4):608-616. doi: 10.1111/j.1939-0025.1979.tb02646.x. PMID 495703
- [Background] Vannatta K, Gartstein MA, Short A, Noll RB. A controlled study of peer relationships of children surviving brain tumors: teacher, peer, and self ratings. J Pediatr Psychol. 1998 Oct;23(5):279-87. doi: 10.1093/jpepsy/23.5.279. PMID 9782676
- [Background] Lavigne JV, Faier-Routman J. Psychological adjustment to pediatric physical disorders: a meta-analytic review. J Pediatr Psychol. 1992 Apr;17(2):133-57. doi: 10.1093/jpepsy/17.2.133. PMID 1534367
- [Background] Patenaude AF, Kupst MJ. Psychosocial functioning in pediatric cancer. J Pediatr Psychol. 2005 Jan-Feb;30(1):9-27. doi: 10.1093/jpepsy/jsi012. PMID 15610981
- [Background] Dolgin MJ, Somer E, Buchvald E, Zaizov R. Quality of life in adult survivors of childhood cancer. Soc Work Health Care. 1999;28(4):31-43. doi: 10.1300/J010v28n04_03. PMID 10425670
- [Background] Oeffinger KC, Robison LL. Childhood cancer survivors, late effects, and a new model for understanding survivorship. JAMA. 2007 Jun 27;297(24):2762-4. doi: 10.1001/jama.297.24.2762. No abstract available. PMID 17595279